CLINICAL TRIAL: NCT06140745
Title: Evaluation of Efficacy of Experimental Dentifrice Formulations With Different Forms of Fluoride and/or Other Agents to Remineralize Enamel and Dentine Subsurface Lesions in a Double-Blind Randomized In-Situ Clinical Trial
Brief Title: Evaluation of Dentifrice Formulations to Remineralize Enamel and Dentine Subsurface Lesions in a Double-Blind In-Situ Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019176
Record Dates: First submitted 2023-11-14; First posted 2023-11-20 (Actual); Last update posted 2023-11-20 (Actual); Status verified 2023-11

CONDITIONS: Caries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 0 ppm Fluoride Dentifrice 1 (Placebo Comparator)
  Interventions: Drug: 0 ppm Fluoride Dentifrice 1
- 1100 ppm NaF Fluoride Dentifrice (Active Comparator)
  Interventions: Drug: 1100 ppm NaF Fluoride Dentifrice
- 1500 ppm NaMFP Fluoride Dentifrice (Active Comparator)
  Interventions: Drug: 1500 ppm NaMFP Fluoride Dentifrice
- 0 ppm Fluoride Dentifrice 2 (Sham Comparator)
  Interventions: Drug: 0 ppm Fluoride Dentifrice 2
- 0 ppm Fluoride Dentifrice 3 (Sham Comparator)
  Interventions: Drug: 0 ppm Fluoride Dentifrice 3

INTERVENTIONS:
Drug: 0 ppm Fluoride Dentifrice 1 — Each subject will use this product during one of the five treatment periods in the crossover study design.
  Arms: 0 ppm Fluoride Dentifrice 1
Drug: 1100 ppm NaF Fluoride Dentifrice — Each subject will use this product during one of the five treatment periods in the crossover study design.
  Arms: 1100 ppm NaF Fluoride Dentifrice
Drug: 1500 ppm NaMFP Fluoride Dentifrice — Each subject will use this product during one of the five treatment periods in the crossover study design.
  Arms: 1500 ppm NaMFP Fluoride Dentifrice
Drug: 0 ppm Fluoride Dentifrice 2 — Each subject will use this product during one of the five treatment periods in the crossover study design.
  Arms: 0 ppm Fluoride Dentifrice 2
Drug: 0 ppm Fluoride Dentifrice 3 — Each subject will use this product during one of the five treatment periods in the crossover study design.
  Arms: 0 ppm Fluoride Dentifrice 3

SUMMARY:
To compare the remineralization and demineralization inhibition potential of early subsurface carious lesions in enamel in situ after rinsing with five different aqueous slurries of toothpaste formulations. Percent remineralization (%R), i.e. the % change in ΔZ values relative to ΔZd, will be the primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Be 18-75 years of age;
* Provide written informed consent prior to participation and be given a signed copy of the informed consent form;
* Be in good general health based on medical/dental history and oral exam;
* Have no history of adverse or allergic reactions to tin or tin-containing products;
* Agree not to participate in any other oral study for the study duration;
* Have a reasonable functional dentition as determined by the oral examiner and sufficient teeth to support the fabricated dental appliance;
* Be willing to participate in the study, able to follow the study directions, successfully tolerate/perform all study procedures, and willing to return for all specified visits at their appointed time;
* Be willing to refrain from using non-study dentifrice, mouth rinse, chewing gum, and other non-study oral care products during the study;
* Be willing to postpone all elective dental procedures until the study has been completed;
* Be willing to refrain from using calcium chews while using the test products;
* Be willing and able to refrain from wearing a nightguard (occlusal splint) for the entire course of the study (for nightguard wearers only).
* Ability to understand, and ability to read and sign, the informed consent form;
* Have at least 22 natural teeth;
* Have a gum-stimulated whole salivary flow rate ≥1.0 ml/minute and unstimulated whole salivary flow rate ≥ 0.2 ml/minute.
* Willingness to comply with all study procedures and be available for the duration of the study.

Exclusion Criteria:

* Advanced periodontal disease, as characterized by purulent exudate, generalized mobility, and/or severe recession;
* Active treatment for periodontitis;
* A medical condition which requires premedication prior to dental visits/procedures;
* Untreated dental problems (e.g. cavities);
* Self-reported pregnancy or plans to become pregnant during the study;
* Existing dental work which prevents wearing of the appliance including orthodontic appliances or removable dentures;
* Chronic disease such as diabetes or use of medications that cause gum swelling;
* Any diseases or conditions (including sensitivity to dentifrice ingredients or a history of allergic or adverse reactions to tin or tin-containing products) that might interfere with examination procedures or the participant safely completing the study;
* Treatment with antibiotics or anti-inflammatory medicines in the month prior to starting the study;
* Use of drugs that may interact with the toothpaste slurries or which may affect salivary flow rate;
* History of health conditions requiring antibiotic coverage prior to dental treatment;
* Serious infectious disease;
* Any other medical or dental conditions deemed to put the health and wellbeing of the participant or research team at risk if the potential participant participated in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-02-21 (Actual); Study Completion 2021-02-21 (Actual)

PRIMARY OUTCOMES:
Mineral Density | 14 days
  The percent mineral profile of each enamel/dentinel slab's demineralized control and remineralized/treated lesion, obtained from the microdensitometry analysis, will be compared with the median sound enamel percent mineral profile of the same section. A negative value indicates mineral has been lost and, therefore, the lesion has progressed, whereas a positive value indicates mineral has been gained and, therefore, the lesion has regressed.
Scanning Electron Microscopy (SEM) | 14 days
  SEM imaging and SEM-EDS analysis will be conducted on TMR sections and whole sections of dentine lesions treated in situ to assess the occlusion of dentine tubules and distribution of elements within the lesions following the experiment.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Melbourne, Melbourne, Australia